CLINICAL TRIAL: NCT04019756
Title: IDENTIFICATION OF URINARY MICROBIOTE IN PATIENTS WITH DIAGNOSTIC-RELATED CYSTOSCOPY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-60; 2018-60 (Registry Identifier: APHM)
Record Dates: First submitted 2019-07-09; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Cystoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cancer: 50 patients ultimately diagnosed with bladder cancer and 50 control patients (diagnosis of cancer reversed at cystoscopy or cystoscopy for another cause)

SUMMARY:
Identify by culture the urinary microbiota of patients with bladder cancer (at the time of diagnosis) and controls.Identify by metagenomics the urinary microbiota of patients with bladder cancer (at the time of diagnosis) and controls.

DETAILED DESCRIPTION:
Relationships between the human microbiota and various pathologies such as cancer have been demonstrated. The microbiota would have an influence on the effectiveness of anticancer treatments.

Bladder cancers are five times more common in men than women, and this difference in incidence has long been explained by a higher smoking rate among men. However, the increase in smoking among women has not led, as in the case of lung cancer, to a significant increase in bladder cancer among them.

Urine bladder has long been considered "sterile" by generations of researchers. Recent studies have shown that most urine is not sterile but instead contains a different microbiota in both men and women. In women Actinobacteria, including Mycobacteria, and Bacteroidetes have been detected.

BCG therapy is used in the treatment of bladder cancer. BCG, in addition to being a vaccine to prevent tuberculosis, is a mycobacterium belonging to the phylum Actinobacteria [4]. Controversial studies have suggested the same potential for Lactobacillus casei. Lactobacillii are Firmicutes found both in the urinary microbiota of men and women.

Thus microbiota composed mainly of Actinobacteria could be associated with a lower incidence of bladder cancers in women.

ELIGIBILITY:
Inclusion Criteria:

* Person receiving a cystoscopy in the context of a suspicion of bladder cancer
* Person and / or legal guardian for minors who have been informed about the study and have not expressed opposition to participate in the study.
* Affiliated person or beneficiary of a social security scheme.

Exclusion Criteria:

* Vulnerable person: pregnant, parturient or nursing woman,
* person under guardianship or curatorship, or deprived of liberty by a judicial or administrative decision.
* Person treated with antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any present patient meeting the inclusion criteria of the study will be offered to participate in the study. For this purpose during the hospitalization or consultation of the patient, the investigator or his collaborator.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-03-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Matrix Assisted Laser Desorption Ionisation - Time of Flight | 1 day
  A matrix and a sample are deposited on a target. Pulsed laser shots desorb the matrix which then ionizes the sample by charge transfer. By potential differences applied to lenses, the ionized molecules are accelerated and then transferred to the TOF analyzer. This analyzer will allow the separation of the ionized molecules which will depend on their mass-to-charge ratio.